CLINICAL TRIAL: NCT05688410
Title: Enhancing Exercise and Psychotherapy to Treat Pain and Addiction in Adults With an Opioid Use Disorder (EXPO): A Randomized Trial (R33 Phase)
Brief Title: Enhancing Exercise and Psychotherapy to Treat Pain and Addiction in Adults With an Opioid Use Disorder (EXPO; R33 Phase)
Acronym: EXPO-R33
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Colorado, Denver (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nora Nock, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20201427 - R33 Phase; 5R33AT010806-03 (NIH)
Record Dates: First submitted 2022-12-23; First posted 2023-01-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2^1 x 3^1 factorial randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Assisted Exercise and I-STOP (Experimental): Participants randomized to "Assisted Exercise" will exercise on a special bike that assists them to pedal faster than they do voluntarily on their own ("assisted" exercise bike). Participants who are randomized to receive I-STOP will receive the "Self-regulation Treatment for Opioid addiction and Pain" (STOP) program modified for inpatients/residential drug treatment (I-STOP).
  Interventions: Other: Exercise; Behavioral: Psychotherapy Pain and Addiction (I-STOP)
- Voluntary Exercise and I-STOP (Experimental): Participants randomized to "Voluntary Exercise" will exercise on a standard stationary bike where they will pedal at their voluntary rates. Participants who are randomized to receive I-STOP will receive the "Self-regulation Treatment for Opioid addiction and Pain" (STOP) program modified for inpatients/residential drug treatment (I-STOP).
  Interventions: Other: Exercise; Behavioral: Psychotherapy Pain and Addiction (I-STOP)
- Assisted Exercise and No I-STOP (Experimental): Participants randomized to "Assisted Exercise" will exercise on a special bike that assists them to pedal faster than they do voluntarily on their own ("assisted" exercise bike). Participants randomized to "No I-STOP" will not receive the psychotherapy for pain and addiction but will receive their standard behavioral treatment as usual (TAU).
  Interventions: Other: Exercise
- Voluntary Exercise and No I-STOP (Experimental): Participants randomized to "Voluntary Exercise" will exercise on a standard stationary bike where they will pedal at their voluntary rates. Participants randomized to "No I-STOP" will not receive the psychotherapy for pain and addiction but will receive their standard behavioral treatment as usual (TAU).
  Interventions: Other: Exercise
- No Exercise and I-STOP (Experimental): Participants randomized to receive "No Exercise" will not receive structured "assisted" or voluntary rate cycling exercise. Participants randomized to "No I-STOP" will not receive the psychotherapy for pain and addiction but will receive their standard behavioral treatment as usual (TAU).
  Interventions: Behavioral: Psychotherapy Pain and Addiction (I-STOP)
- No Exercise and No I-STOP (No Intervention): Participants randomized to receive "No Exercise" will not receive structured "assisted" or voluntary rate cycling exercise. Participants randomized to "No I-STOP" will not receive the psychotherapy for pain and addiction but will receive their standard behavioral treatment as usual (TAU).

INTERVENTIONS:
Other: Exercise — Participants who are randomized to exercise will be perform exercise on stationary bikes. Participants randomized to "Voluntary Exercise" will exercise on a standard stationary bike where they will pedal at their voluntary rates. Participants randomized to "Assisted Exercise" will exercise on a special bike that assists them to pedal faster than they do voluntarily on their own ("assisted (exercise) bike").
  Arms: Assisted Exercise and I-STOP; Assisted Exercise and No I-STOP; Voluntary Exercise and I-STOP; Voluntary Exercise and No I-STOP
Behavioral: Psychotherapy Pain and Addiction (I-STOP) — Participants who are randomized to receive I-STOP will receive the "Self-regulation Treatment for Opioid addiction and Pain" (STOP) program modified for inpatients/residential drug treatment (I-STOP). I-STOP uses empirically validated pain psychotherapy approaches targeted to patients with an OUD using psycho-physiological self-regulation components and biofeedback with "Bio-dots".
  Arms: Assisted Exercise and I-STOP; No Exercise and I-STOP; Voluntary Exercise and I-STOP

SUMMARY:
This work will involve conducting a randomized trial that will evaluate preliminary efficacy of "assisted" rate cycling, voluntary rate cycling and psychotherapy for pain individually and in combination as adjunctive treatments on cravings (primary outcome) in adults with an opioid use disorder. The investigators will also evaluate the effects of "assisted" rate cycling, voluntary rate cycling and I-STOP on secondary outcomes including depression, anxiety and sleep.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Must be enrolled in a residential/inpatient drug treatment program at a collaborating drug treatment center
* Must be diagnosed with an Opioid Use Disorder (OUD; ICD-10 F11.20) or a Poly-substance Drug Use that includes an opioid component (ICD-10,F19.xx)
* Must have self-reported pain or a pain condition describing a non-cancer related chronic pain disorder
* Must be approved to exercise in the study by the drug treatment center (Medical Director, physician or other relevant clinical staff or primary care physician (PCP))

Exclusion Criteria:

* Any substantive contraindications to exercise
* Psychiatrically unstable
* Pregnant women
* Non-English speaking adults
* Adults unable to provide informed written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Drug cravings | Change from baseline to intervention program completion, an average of 8 weeks
  Change in drug cravings: self-report, visual analog scale (VAS), higher scores indicate higher levels of cravings;

SECONDARY OUTCOMES:
Depression | Change from baseline to intervention program completion, an average of 8 weeks
  Change in depression: self-report, standardized questionnaire (Depression sub-scale in Hospital Anxiety and Depression Scale, HADS); Total Score range: 0-21; higher scores indicate higher levels of depression
Anxiety | Change from baseline to intervention program completion, an average of 8 weeks
  Change in anxiety: self-report, standardized questionnaire (Depression sub-scale in Hospital Anxiety and Depression Scale, HADS); Total Score range: 0-21; Higher scores indicate higher levels of anxiety
Sleep | Change from baseline to intervention program completion, an average of 8 weeks
  Change in sleep: self-report, standardized questionnaire (Pittsburgh Sleep Quality Index, PSQI); Total Score range: 0-21; Higher scores indicate poorer sleep quality
Drug Cravings using Questionnaire | Change from baseline to intervention program completion, an average of 8 weeks
  standardized questionnaire (Desires for Drug Questionnaire), higher scores indicate higher levels of cravings

CONTACTS AND LOCATIONS:
Overall Officials: Nora L. Nock, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - University of Colorado at Denver, Denver, Colorado
  - Case Western Reserve University, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared as required by NIH HEAL and as deemed acceptable by governing IRB, HIPPA and other regulations.